CLINICAL TRIAL: NCT00504413
Title: Role of CYP2B6, CYP3A4, and MDR1 in the Metabolic Clearance of Methadone in Human Subjects
Brief Title: Role of CYP2B6, CYP3A4, and MDR1 in the Metabolic Clearance of Methadone
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Rheem Totah/Assistant Professor, Medicinal Chemistry, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 30931-A; 06-3659-A 01
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Substance-Related Disorders
Keywords: Metabolic Networks and Pathways; Methadone; Polymorphism, genetic; Cytochrome P-450 Enzyme System
MeSH Terms: conditions — Substance-Related Disorders | interventions — Digoxin; Pharmaceutical Preparations; Bupropion; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: midazolam(drug), digoxin (drug) — Midazolam (2mg po) and digoxin (0.5mg po) will be administered one time, an hour apart. Blood concentration will be collected at various points in an 8 hour period.
Drug: Bupropion (drug) — Bupropion (150mg po) will be administered one time on a separate visit. Blood concentrations will be collected at various points in a 72 hour period.
  Other Names: Wellbutrin
Drug: Methadone (drug) — Methadone (10mg po) will be administered at a separate visit 2 weeks after the bupropion visit. The dose is given once. Blood concentrations will be measured at various points in a 72 hour period. Pupil constriction will be measured and urine will be collected during this period as well.

SUMMARY:
The purpose of this study is to determine to what extent CYP2B6, CYP3A4, and MDR1 polymorphisms affect the metabolism of methadone.

DETAILED DESCRIPTION:
Methadone maintenance treatment (MMT) has been used to rehabilitate the opiate addict resulting in a higher quality of life for the patient as well as improving social and psychological functioning while reducing the overall cost to society. The maintenance dose of methadone is highly variable between patients, and drug-drug interactions have been observed between methadone and various medications used to treat a variety of diseases. Identification and understanding of the enzymes responsible for the metabolism of methadone could potentially lead to improved strategy in individualizing methadone dosing and reduce the risk of adverse drug interactions.

Several cytochrome P450 enzymes (CYPs) have been identified and hypothesized to be involved in methadone metabolism in vitro, particularly CYP2B6 and CYP3A4. However, the quantitative contribution of CYP2B6 and CYP3A4 in the elimination clearance of methadone in vivo remains undefined. In addition, methadone is a substrate of the efflux transporter, P-glycoprotein (Pgp) at the intestinal mucosa. We are proposing a pilot study in healthy human subjects to investigate the following hypotheses:

1. Pgp limits the gastrointestinal absorption
2. Inter-subject variations in CYP2B6 and CYP3A4 activities explain the variation in methadone clearance in vivo

This will be accomplished by correlating the pharmacokinetics of methadone and the phenotype probes for Pgp (digoxin), CYP2B6 (bupropion) and CYP3A4 (midazolam). We plan to use these data to design a human subject study to assess the utility of MDR1 and CYP genotyping in predicting the methadone maintenance dose in a cohort of MMT patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Within 25% of ideal body weight

Exclusion Criteria:

* Pregnant
* A prisoner
* Enemy, non-combatant
* Smoker
* Have a history of liver disease
* Have a history of heart disease
* Have a history of drug abuse
* Currently on prescription medication

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-07; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Explore if there is a correlation between the areas of the concentration curves of probe substrates for CYP3A4 and/or CYP2B6 and Pgp and the area of the concentration curve of methadone. | two years

SECONDARY OUTCOMES:
LC-MS assays will be developed to analyze the plasma content of the probe substrates, methadone and their metabolites. Specifically, midazolam, 1-OH midazolam, bupropion, t-butyl-hydroxy bupropion, digoxin, methadone, and EDDP (a methadone metabolite). | two years
Isolate and bank the DNA of the subjects for future genotyping of variant alleles that will be identified in this study to be important in methadone pharmacokinetics. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Rheem A Totah, PhD, Principal Investigator — University of Washington, Medicinal Chemistry Department
Locations (1):
- University of Washington General Clinical Research Center, Seattle, Washington, United States

REFERENCES:
- [Background] Beckett AH, Taylor JF, Casy AF, Hassan MM. The biotransformation of methadone in man: synthesis and identification of a major metabolite. J Pharm Pharmacol. 1968 Oct;20(10):754-62. doi: 10.1111/j.2042-7158.1968.tb09634.x. No abstract available. PMID 4386743
- [Background] Kreek MJ, Vocci FJ. History and current status of opioid maintenance treatments: blending conference session. J Subst Abuse Treat. 2002 Sep;23(2):93-105. doi: 10.1016/s0740-5472(02)00259-3. PMID 12220607
- [Background] Mattick RP, Breen C, Kimber J, Davoli M. Methadone maintenance therapy versus no opioid replacement therapy for opioid dependence. Cochrane Database Syst Rev. 2003;(2):CD002209. doi: 10.1002/14651858.CD002209. PMID 12804430
- [Background] Brettle RP. HIV and harm reduction for injection drug users. AIDS. 1991 Feb;5(2):125-36. doi: 10.1097/00002030-199102000-00001. No abstract available. PMID 2031687
- [Background] Ward J, Mattrick R, Hall W. Methadone maintenance treatment and other opioid replacement therapies. Harwood Academic Publishers, Amsterdam. 1998
- [Background] Caplehorn JR, Drummer OH. Mortality associated with New South Wales methadone programs in 1994: lives lost and saved. Med J Aust. 1999 Feb 1;170(3):104-9. doi: 10.5694/j.1326-5377.1999.tb127675.x. PMID 10065120
- [Background] Sorensen JL, Copeland AL. Drug abuse treatment as an HIV prevention strategy: a review. Drug Alcohol Depend. 2000 Apr 1;59(1):17-31. doi: 10.1016/s0376-8716(99)00104-0. PMID 10706972
- [Background] Stenbacka M, Leifman A, Romelsjo A. The impact of methadone treatment on registered convictions and arrests in HIV-positive and HIV-negative men and women with one or more treatment periods. Drug Alcohol Rev. 2003 Mar;22(1):27-34. doi: 10.1080/0959523021000059802. PMID 12745356
- [Background] Wong KH, Lee SS, Lim WL, Low HK. Adherence to methadone is associated with a lower level of HIV-related risk behaviors in drug users. J Subst Abuse Treat. 2003 Apr;24(3):233-9. doi: 10.1016/s0740-5472(03)00029-1. PMID 12810144
- [Background] Bruera E, Kim HN. Cancer pain. JAMA. 2003 Nov 12;290(18):2476-9. doi: 10.1001/jama.290.18.2476. No abstract available. PMID 14612485
- [Background] Gourlay GK, Cherry DA, Cousins MJ. A comparative study of the efficacy and pharmacokinetics of oral methadone and morphine in the treatment of severe pain in patients with cancer. Pain. 1986 Jun;25(3):297-312. doi: 10.1016/0304-3959(86)90234-4. PMID 3528988
- [Background] Manfredi PL, Borsook D, Chandler SW, Payne R. Intravenous methadone for cancer pain unrelieved by morphine and hydromorphone: clinical observations. Pain. 1997 Mar;70(1):99-101. doi: 10.1016/s0304-3959(96)03313-1. PMID 9106815
- [Background] Mercadante S. Methadone in cancer pain. Eur J Pain. 1997;1(2):77-83; discussion 84-5. doi: 10.1016/s1090-3801(97)90064-1. PMID 15102407
- [Background] Ripamonti C, Bianchi M. The use of methadone for cancer pain. Hematol Oncol Clin North Am. 2002 Jun;16(3):543-55. doi: 10.1016/s0889-8588(02)00017-5. PMID 12170567
- [Background] Kristensen K, Christensen CB, Christrup LL. The mu1, mu2, delta, kappa opioid receptor binding profiles of methadone stereoisomers and morphine. Life Sci. 1995;56(2):PL45-50. doi: 10.1016/0024-3205(94)00426-s. PMID 7823756
- [Background] Begre S, von Bardeleben U, Ladewig D, Jaquet-Rochat S, Cosendai-Savary L, Golay KP, Kosel M, Baumann P, Eap CB. Paroxetine increases steady-state concentrations of (R)-methadone in CYP2D6 extensive but not poor metabolizers. J Clin Psychopharmacol. 2002 Apr;22(2):211-5. doi: 10.1097/00004714-200204000-00017. PMID 11910269
- [Background] Inturrisi CE, Verebely K. Disposition of methadone in man after a single oral dose. Clin Pharmacol Ther. 1972 Nov-Dec;13(6):923-30. doi: 10.1002/cpt1972136923. No abstract available. PMID 5081605
- [Background] Hanna J, Foster DJ, Salter A, Somogyi AA, White JM, Bochner F. Within- and between- subject variability in methadone pharmacokinetics and pharmacodynamics in methadone maintenance subjects. Br J Clin Pharmacol. 2005 Oct;60(4):404-13. doi: 10.1111/j.1365-2125.2005.02464.x. PMID 16187972
- [Background] Peles E, Schreiber S, Gordon J, Adelson M. Significantly higher methadone dose for methadone maintenance treatment (MMT) patients with chronic pain. Pain. 2005 Feb;113(3):340-346. doi: 10.1016/j.pain.2004.11.011. PMID 15661442
- [Background] Charlier C, Dessalles MC, Plomteux G. Methadone maintenance treatment: is it possible to adapt the daily doses to the metabolic activity of the patient? Ther Drug Monit. 2001 Feb;23(1):1-3. doi: 10.1097/00007691-200102000-00001. PMID 11206036
- [Background] Shinderman M, Maxwell S, Brawand-Amey M, Golay KP, Baumann P, Eap CB. Cytochrome P4503A4 metabolic activity, methadone blood concentrations, and methadone doses. Drug Alcohol Depend. 2003 Mar 1;69(2):205-11. doi: 10.1016/s0376-8716(02)00320-4. PMID 12609702
- [Background] Eap CB, Buclin T, Baumann P. Interindividual variability of the clinical pharmacokinetics of methadone: implications for the treatment of opioid dependence. Clin Pharmacokinet. 2002;41(14):1153-93. doi: 10.2165/00003088-200241140-00003. PMID 12405865
- [Background] Foster DJ, Somogyi AA, Dyer KR, White JM, Bochner F. Steady-state pharmacokinetics of (R)- and (S)-methadone in methadone maintenance patients. Br J Clin Pharmacol. 2000 Nov;50(5):427-40. doi: 10.1046/j.1365-2125.2000.00272.x. PMID 11069437
- [Background] Iribarne C, Dreano Y, Bardou LG, Menez JF, Berthou F. Interaction of methadone with substrates of human hepatic cytochrome P450 3A4. Toxicology. 1997 Feb 14;117(1):13-23. doi: 10.1016/s0300-483x(96)03549-4. PMID 9020195
- [Background] Niemi M, Backman JT, Fromm MF, Neuvonen PJ, Kivisto KT. Pharmacokinetic interactions with rifampicin : clinical relevance. Clin Pharmacokinet. 2003;42(9):819-50. doi: 10.2165/00003088-200342090-00003. PMID 12882588
- [Background] Gerber JG, Rhodes RJ, Gal J. Stereoselective metabolism of methadone N-demethylation by cytochrome P4502B6 and 2C19. Chirality. 2004 Jan;16(1):36-44. doi: 10.1002/chir.10303. PMID 14628297
- [Background] Kharasch ED, Hoffer C, Whittington D, Sheffels P. Role of hepatic and intestinal cytochrome P450 3A and 2B6 in the metabolism, disposition, and miotic effects of methadone. Clin Pharmacol Ther. 2004 Sep;76(3):250-69. doi: 10.1016/j.clpt.2004.05.003. PMID 15371986
- [Background] Moody DE, Walsh SL, Rollins DE, Neff JA, Huang W. Ketoconazole, a cytochrome P450 3A4 inhibitor, markedly increases concentrations of levo-acetyl-alpha-methadol in opioid-naive individuals. Clin Pharmacol Ther. 2004 Aug;76(2):154-66. doi: 10.1016/j.clpt.2004.04.004. PMID 15289792
- [Background] Oda Y, Kharasch ED. Metabolism of methadone and levo-alpha-acetylmethadol (LAAM) by human intestinal cytochrome P450 3A4 (CYP3A4): potential contribution of intestinal metabolism to presystemic clearance and bioactivation. J Pharmacol Exp Ther. 2001 Sep;298(3):1021-32. PMID 11504799
- [Background] Wang JS, DeVane CL. Involvement of CYP3A4, CYP2C8, and CYP2D6 in the metabolism of (R)- and (S)-methadone in vitro. Drug Metab Dispos. 2003 Jun;31(6):742-7. doi: 10.1124/dmd.31.6.742. PMID 12756206
- [Background] Boulton DW, Arnaud P, DeVane CL. Pharmacokinetics and pharmacodynamics of methadone enantiomers after a single oral dose of racemate. Clin Pharmacol Ther. 2001 Jul;70(1):48-57. doi: 10.1067/mcp.2001.116793. PMID 11452244
- [Background] Faucette SR, Wang H, Hamilton GA, Jolley SL, Gilbert D, Lindley C, Yan B, Negishi M, LeCluyse EL. Regulation of CYP2B6 in primary human hepatocytes by prototypical inducers. Drug Metab Dispos. 2004 Mar;32(3):348-58. doi: 10.1124/dmd.32.3.348. PMID 14977870
- [Background] Hesse LM, Sakai Y, Vishnuvardhan D, Li AP, von Moltke LL, Greenblatt DJ. Effect of bupropion on CYP2B6 and CYP3A4 catalytic activity, immunoreactive protein and mRNA levels in primary human hepatocytes: comparison with rifampicin. J Pharm Pharmacol. 2003 Sep;55(9):1229-39. doi: 10.1211/0022357021657. PMID 14604466
- [Background] Martin H, Sarsat JP, de Waziers I, Housset C, Balladur P, Beaune P, Albaladejo V, Lerche-Langrand C. Induction of cytochrome P450 2B6 and 3A4 expression by phenobarbital and cyclophosphamide in cultured human liver slices. Pharm Res. 2003 Apr;20(4):557-68. doi: 10.1023/a:1023234429596. PMID 12739762
- [Background] Parkinson A, Mudra DR, Johnson C, Dwyer A, Carroll KM. The effects of gender, age, ethnicity, and liver cirrhosis on cytochrome P450 enzyme activity in human liver microsomes and inducibility in cultured human hepatocytes. Toxicol Appl Pharmacol. 2004 Sep 15;199(3):193-209. doi: 10.1016/j.taap.2004.01.010. PMID 15364537
- [Background] Pascussi JM, Gerbal-Chaloin S, Drocourt L, Maurel P, Vilarem MJ. The expression of CYP2B6, CYP2C9 and CYP3A4 genes: a tangle of networks of nuclear and steroid receptors. Biochim Biophys Acta. 2003 Feb 17;1619(3):243-53. doi: 10.1016/s0304-4165(02)00483-x. PMID 12573484
- [Background] Crettol S, Deglon JJ, Besson J, Croquette-Krokkar M, Gothuey I, Hammig R, Monnat M, Huttemann H, Baumann P, Eap CB. Methadone enantiomer plasma levels, CYP2B6, CYP2C19, and CYP2C9 genotypes, and response to treatment. Clin Pharmacol Ther. 2005 Dec;78(6):593-604. doi: 10.1016/j.clpt.2005.08.011. PMID 16338275
- [Background] Lotsch J, Skarke C, Wieting J, Oertel BG, Schmidt H, Brockmoller J, Geisslinger G. Modulation of the central nervous effects of levomethadone by genetic polymorphisms potentially affecting its metabolism, distribution, and drug action. Clin Pharmacol Ther. 2006 Jan;79(1):72-89. doi: 10.1016/j.clpt.2005.09.010. PMID 16413243
- [Background] Miksys S, Lerman C, Shields PG, Mash DC, Tyndale RF. Smoking, alcoholism and genetic polymorphisms alter CYP2B6 levels in human brain. Neuropharmacology. 2003 Jul;45(1):122-32. doi: 10.1016/s0028-3908(03)00136-9. PMID 12814665
- [Background] Pelkonen O, Maenpaa J, Taavitsainen P, Rautio A, Raunio H. Inhibition and induction of human cytochrome P450 (CYP) enzymes. Xenobiotica. 1998 Dec;28(12):1203-53. doi: 10.1080/004982598238886. No abstract available. PMID 9890159
- [Background] de Boer AG, van der Sandt IC, Gaillard PJ. The role of drug transporters at the blood-brain barrier. Annu Rev Pharmacol Toxicol. 2003;43:629-56. doi: 10.1146/annurev.pharmtox.43.100901.140204. Epub 2002 Jan 10. PMID 12415123
- [Background] Fricker G, Miller DS. Relevance of multidrug resistance proteins for intestinal drug absorption in vitro and in vivo. Pharmacol Toxicol. 2002 Jan;90(1):5-13. doi: 10.1034/j.1600-0773.2002.900103.x. PMID 12005113
- [Background] Fromm MF. P-glycoprotein: a defense mechanism limiting oral bioavailability and CNS accumulation of drugs. Int J Clin Pharmacol Ther. 2000 Feb;38(2):69-74. doi: 10.5414/cpp38069. PMID 10706193
- [Background] Lamba J, Strom S, Venkataramanan R, Thummel KE, Lin YS, Liu W, Cheng C, Lamba V, Watkins PB, Schuetz E. MDR1 genotype is associated with hepatic cytochrome P450 3A4 basal and induction phenotype. Clin Pharmacol Ther. 2006 Apr;79(4):325-38. doi: 10.1016/j.clpt.2005.11.013. Epub 2006 Feb 20. PMID 16580901
- [Background] Lin JH, Yamazaki M. Role of P-glycoprotein in pharmacokinetics: clinical implications. Clin Pharmacokinet. 2003;42(1):59-98. doi: 10.2165/00003088-200342010-00003. PMID 12489979
- [Background] Bouer R, Barthe L, Philibert C, Tournaire C, Woodley J, Houin G. The roles of P-glycoprotein and intracellular metabolism in the intestinal absorption of methadone: in vitro studies using the rat everted intestinal sac. Fundam Clin Pharmacol. 1999;13(4):494-500. doi: 10.1111/j.1472-8206.1999.tb00009.x. PMID 10456292
- [Background] Callaghan R, Riordan JR. Synthetic and natural opiates interact with P-glycoprotein in multidrug-resistant cells. J Biol Chem. 1993 Jul 25;268(21):16059-64. PMID 8101846
- [Background] Stormer E, Perloff MD, von Moltke LL, Greenblatt DJ. Methadone inhibits rhodamine123 transport in Caco-2 cells. Drug Metab Dispos. 2001 Jul;29(7):954-6. PMID 11408360
- [Background] Thompson SJ, Koszdin K, Bernards CM. Opiate-induced analgesia is increased and prolonged in mice lacking P-glycoprotein. Anesthesiology. 2000 May;92(5):1392-9. doi: 10.1097/00000542-200005000-00030. PMID 10781286
- [Background] Kharasch ED, Hoffer C, Whittington D. The effect of quinidine, used as a probe for the involvement of P-glycoprotein, on the intestinal absorption and pharmacodynamics of methadone. Br J Clin Pharmacol. 2004 May;57(5):600-10. doi: 10.1111/j.1365-2125.2003.02053.x. PMID 15089813
- [Background] Wang JS, Ruan Y, Taylor RM, Donovan JL, Markowitz JS, DeVane CL. Brain penetration of methadone (R)- and (S)-enantiomers is greatly increased by P-glycoprotein deficiency in the blood-brain barrier of Abcb1a gene knockout mice. Psychopharmacology (Berl). 2004 Apr;173(1-2):132-8. doi: 10.1007/s00213-003-1718-1. Epub 2004 Jan 8. PMID 14712343
- [Background] Streetman DS, Bertino JS Jr, Nafziger AN. Phenotyping of drug-metabolizing enzymes in adults: a review of in-vivo cytochrome P450 phenotyping probes. Pharmacogenetics. 2000 Apr;10(3):187-216. doi: 10.1097/00008571-200004000-00001. PMID 10803676
- [Background] Streetman DS, Bleakley JF, Kim JS, Nafziger AN, Leeder JS, Gaedigk A, Gotschall R, Kearns GL, Bertino JS Jr. Combined phenotypic assessment of CYP1A2, CYP2C19, CYP2D6, CYP3A, N-acetyltransferase-2, and xanthine oxidase with the "Cooperstown cocktail". Clin Pharmacol Ther. 2000 Oct;68(4):375-83. doi: 10.1067/mcp.2000.109519. PMID 11061577
- [Background] Doherty JE, Flanigan WJ, Murphy ML, Bulloch RT, Dalrymple GL, Beard OW, Perkins WH. Tritiated digoxin. XIV. Enterohepatic circulation, absorption, and excretion studies in human volunteers. Circulation. 1970 Nov;42(5):867-73. doi: 10.1161/01.cir.42.5.867. No abstract available. PMID 5477259
- [Background] Klotz U, Antonin KH. Biliary excretion studies with digoxin in man. Int J Clin Pharmacol Biopharm. 1977 Jul;15(7):332-4. PMID 892949
- [Background] Palovaara S, Pelkonen O, Uusitalo J, Lundgren S, Laine K. Inhibition of cytochrome P450 2B6 activity by hormone replacement therapy and oral contraceptive as measured by bupropion hydroxylation. Clin Pharmacol Ther. 2003 Oct;74(4):326-33. doi: 10.1016/S0009-9236(03)00202-9. PMID 14534519
- [Background] Turpeinen M, Nieminen R, Juntunen T, Taavitsainen P, Raunio H, Pelkonen O. Selective inhibition of CYP2B6-catalyzed bupropion hydroxylation in human liver microsomes in vitro. Drug Metab Dispos. 2004 Jun;32(6):626-31. doi: 10.1124/dmd.32.6.626. PMID 15155554
- [Background] Rosner B. Fundamentals of Biostatistics. Duxbury, 2006.
- [Background] Whittington D, Sheffels P, Kharasch ED. Stereoselective determination of methadone and the primary metabolite EDDP in human plasma by automated on-line extraction and liquid chromatography mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2004 Oct 5;809(2):313-21. doi: 10.1016/j.jchromb.2004.06.041. PMID 15315782
- [Background] Jabor VA, Coelho EB, Dos Santos NA, Bonato PS, Lanchote VL. A highly sensitive LC-MS-MS assay for analysis of midazolam and its major metabolite in human plasma: applications to drug metabolism. J Chromatogr B Analyt Technol Biomed Life Sci. 2005 Aug 5;822(1-2):27-32. doi: 10.1016/j.jchromb.2005.05.011. PMID 15993663
- [Background] Tracqui A, Kintz P, Ludes B, Mangin P. High-performance liquid chromatography-ionspray mass spectrometry for the specific determination of digoxin and some related cardiac glycosides in human plasma. J Chromatogr B Biomed Sci Appl. 1997 Apr 25;692(1):101-9. doi: 10.1016/s0378-4347(96)00462-8. PMID 9187389
- [Background] Hsyu PH, Singh A, Giargiari TD, Dunn JA, Ascher JA, Johnston JA. Pharmacokinetics of bupropion and its metabolites in cigarette smokers versus nonsmokers. J Clin Pharmacol. 1997 Aug;37(8):737-43. doi: 10.1002/j.1552-4604.1997.tb04361.x. PMID 9378846
- [Background] Allen DM. The prediction sum of squares as a criterion for selecting predictor variables. In University of Ky Dept of Statistics Tech Report 23, 1971